CLINICAL TRIAL: NCT06156202
Title: Evaluating a Comprehensive Multimodal Outpatient Rehabilitation Program to Improve the Functioning of Persons Suffering From Post-acute Sequelae of SARS-CoV-2 Infection (PASC): A Randomized Controlled
Brief Title: Evaluating a Comprehensive Multimodal Outpatient Rehabilitation Program for PASC Program to Improve Functioning of Persons Suffering From Post-COVID-19 Syndrome: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Medical College of Wisconsin (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 853695
Record Dates: First submitted 2023-11-28; First posted 2023-12-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Post-Acute COVID-19; Post-Acute COVID-19 Syndrome; Post-Acute COVID-19 Infection; Long COVID; Long Covid19; Dyspnea; Orthostasis; Cognitive Impairment
Keywords: PASC; Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; Dyspnea; Dizziness; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented Usual Care (Active Comparator): Following randomization, subjects in the augmented usual care group will be given the results of their in-person baseline assessment as well as the WHO Guide "Support for Rehabilitation Self-Management after COVID-19 Related Illness." This guide consists of ways to manage: breathlessness, difficulty with voice, eating, drinking and swallowing; problems with attention, memory and thinking clearly; limitations in activities of daily living, manage stress and mood dysfunction and advice for when to contact healthcare professionals. Follow-up interviews will assess process measures, including use of outpatient rehabilitation clinics, to examine possible contamination effects
  Interventions: Other: Augmented Usual Care
- Comprehensive Rehabilitation (Experimental): Subjects will be given the option to undergo the comprehensive rehabilitation program including speech therapy and physical therapy. Progression through the rehabilitation program will be personalized and designed based on impairments identified during the comprehensive baseline assessment and previous sessions. Subjects will undergo 12 one- hour sessions over the course of six weeks. The exercise program will be graded and targeted to the person's physical capacity with the goal of slowly advancing the exercise duration or intensity to effect physiological strengthening and increased physical function.
  Interventions: Other: Comprehensive Rehabilitation

INTERVENTIONS:
Other: Comprehensive Rehabilitation — Subjects will be given the option to undergo the comprehensive rehabilitation program including speech therapy and physical therapy. Progression through the rehabilitation program will be personalized and designed based on impairments identified during the comprehensive baseline assessment and previous sessions. Subjects will undergo 12 one- hour sessions over the course of six weeks. The exercise program will be graded and targeted to the person's physical capacity with the goal of slowly advancing the exercise duration or intensity to effect physiological strengthening and increased physical function.
  Arms: Comprehensive Rehabilitation
Other: Augmented Usual Care — Following randomization, subjects in the augmented usual care group will be given the results of their in-person baseline assessment as well as the WHO Guide "Support for Rehabilitation Self-Management after COVID-19 Related Illness." This guide consists of ways to manage: breathlessness, difficulty with voice, eating, drinking and swallowing; problems with attention, memory and thinking clearly; limitations in activities of daily living, manage stress and mood dysfunction and advice for when to contact healthcare professionals. Follow-up interviews will assess process measures, including use of outpatient rehabilitation clinics, to examine possible contamination effects
  Arms: Augmented Usual Care

SUMMARY:
About 10-20% of persons who contract SARS CoV-2 will experience persistent post-acute sequelae of SARSCoV-2 infection (referred here as PASC). While treatments offered at emerging outpatient COVID recovery clinics are being informed by previous similar diseases, the need is great for a better understanding of the unique needs of this growing population and for tested, efficacious rehabilitation programs to address them. We provide both here.The targeted six-week program will be comprised of a core set of therapies, including individually titrated stretching and flexibility, strengthening of accessory breathing muscles and diaphragm, resistance and aerobic conditioning, and vestibular rehabilitation, supplemented by neuropsychological and cognitive remediation tailored to patients' needs.

DETAILED DESCRIPTION:
About 10-20% of persons who contract SARS CoV-2 will experience persistent post-acute sequelae of SARSCoV-2 infection (referred here as PASC). Given that persistent symptoms are heterogeneous with multisystem involvement, recent consensus recommendations suggest that a holistic rehabilitation program may be required to manage PASC and restore function. While treatments offered at emerging outpatient COVID recovery clinics are being informed by previous similar diseases, the need is great for a better understanding of the unique needs of this growing population and for tested, efficacious rehabilitation programs to address them. We provide both here. Specifically, our aims are: (1) To quantify the incidence and severity of PASC across different variants and their effects on health and functioning; (2) To develop and evaluate the effectiveness of a patient-centered, interdisciplinary, multimodal comprehensive rehabilitation program among patients with PASC; and (3)To estimate the costs associated with the proposed PASC rehabilitation intervention and to examine the relationship between intervention's costs and effectiveness and their implication for rehabilitation program initiatives. Data from a large and diverse ongoing longitudinal survey of persons who tested for COVID-19 at the study health system will serve as the sampling frame from which to identify and enroll PASC patients in the study. The targeted six-week program will be comprised of a core set of therapies, including individually titrated stretching and flexibility, strengthening of accessory breathing muscles and diaphragm, resistance and aerobic conditioning, and vestibular rehabilitation, supplemented by neuropsychological and cognitive remediation tailored to patients' needs. Using a randomized controlled trial (RCT) design, the effectiveness of the intervention will be compared to that of usual care augmented by a onetime in-person assessment and patient education materials. In addition to walking speed, a widely used global measure of aerobic capacity and endurance, and patient-reported health and functioning (primary outcomes), we will assess the intervention effectiveness on: (i) cognitive functioning, (ii) pain, (iii) fatigue, (iv) tension, stress, anxiety, and depression, and (v) self-management of PASC symptoms (secondary outcomes). Outcomes will be measured at fixed points in time at 8 weeks (shortly after therapy completion) and at 90 day's post- study entry to examine sustainability of effects. Our overarching hypothesis is that that higher intervention costs in the intervention group will be more than offset by greater improvements in outcomes implying that, overall, persons in the intervention group will receive more cost-effective care than those in usual care group. Given the dearth of rigorous scientific evidence regarding effective assessment and treatment of PASC and the unresolved questions concerning access to and value of post-COVID rehabilitation care, the results of this study will have significant implications for both policy and program development.

ELIGIBILITY:
Inclusion Criteria:

* 18 years if age or older
* English or Spanish speaking
* Previously tested positive for COVID
* Still having symptoms not explained by any other etiologies
* Cognitive impairment
* Fatigue

Exclusion Criteria:

* Participation in another clinical trial
* Score greater than 12 on the fatigue scale
* Score greater than 30 on the memory/thinking scale
* Severe cognitive impairment (i.e. Alzheimer's, Dementia)
* Mental or physical inability to participate in the program

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Six minute walk test | At week 1 and week 8

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dillingham, MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pezzin LE, Larson ER, Lorber W, McGinley EL, Dillingham TR. Music-instruction intervention for treatment of post-traumatic stress disorder: a randomized pilot study. BMC Psychol. 2018 Dec 19;6(1):60. doi: 10.1186/s40359-018-0274-8. PMID 30567598
- [Background] Abramoff BA, Dillingham TR, Caldera FE, Ritchie MD, Pezzin LE. Inpatient Rehabilitation Outcomes After Severe COVID-19 Infections: A Retrospective Cohort Study. Am J Phys Med Rehabil. 2021 Dec 1;100(12):1109-1114. doi: 10.1097/PHM.0000000000001885. PMID 34657085
- [Background] Dillingham T, Kenia J, Shofer F, Marschalek J. A Prospective Assessment of an Adjustable, Immediate Fit, Transtibial Prosthesis. PM R. 2019 Nov;11(11):1210-1217. doi: 10.1002/pmrj.12133. Epub 2019 Apr 1. PMID 30734517
- [Background] McCloskey C, Kenia J, Shofer F, Marschalek J, Dillingham T. Improved Self-Reported Comfort, Stability, and Limb Temperature Regulation with an Immediate Fit, Adjustable Transtibial Prosthesis. Arch Rehabil Res Clin Transl. 2020 Dec;2(4):100090. doi: 10.1016/j.arrct.2020.100090. Epub 2020 Nov 2. PMID 33381750
- [Derived] Abramoff B, Dillingham T, Rybicki AK, Shofer F, McGinley E, Verma SS, Kuns MC, Barry JT, Pezzin LE. Evaluating a Comprehensive Multimodal Outpatient Rehabilitation Program to Improve the Functioning of Persons Suffering from Post-acute Sequelae of SARS-CoV-2 infection (PASC): A Randomized Controlled Trial. Res Sq [Preprint]. 2025 Aug 18:rs.3.rs-7375832. doi: 10.21203/rs.3.rs-7375832/v1. PMID 40894014

DOCUMENTS (1):
  • Informed Consent Form (2023-10-20): https://cdn.clinicaltrials.gov/large-docs/02/NCT06156202/ICF_000.pdf